CLINICAL TRIAL: NCT01570829
Title: Multicentric Double-blind Placebo-controlled Randomized Parallel-group Clinical Trial of Safety and Efficacy of New Dosage Schedule for Dietressa Drug in Treatment of Obese Patients
Brief Title: Clinical Trial of Safety and Efficacy of New Dosage Schedule for Dietressa Drug in Treatment of Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-DI-003
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2019-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Dietressa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietressa (Experimental): Tablet for oral use. 1 tablet 6 times a day. The duration of Dietressa therapy is 24 weeks.
  Interventions: Drug: Dietressa
- Placebo (Placebo Comparator): Tablet for oral use. 1 tablet 6 times a day. The duration of Placebo therapy is 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dietressa — Oral administration.
  Arms: Dietressa
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
* To assess safety of Dietressa in the dose of 6 tablets daily within 24 weeks in treatment of obese patients (BMI 35,0-39,9 kg/m2).
* To assess clinical efficacy of Dietressa in the dose of 6 tablets daily after 24 weeks of therapy in reducing body weight in obese patients (BMI 35,0-39,9 kg/m2).

DETAILED DESCRIPTION:
In general, patients will be observed during 24 weeks of trial.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient subjects with BMI 35,0-39,9 kg/m2.
2. Males or females aged from 18 to 65 years.
3. Use of and compliance with contraception methods by patients of reproductive age, of both sexes.
4. Presence of the patient's information sheet (informed consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Symptomatic (secondary) obesity:

   * with established genetic defect (including as a part of known genetic syndromes affecting multiple organs): Prader-Willi syndrome, Alstrom's syndrome, Laurence-Moon-Biedl syndrome, Dercum's syndrome etc.
   * cerebral (adiposogenital dystrophy, Babinski-Frohlich syndrome): brain tumors; dissemination of systemic lesions, infectious diseases; against mental diseases.
   * endocrine: hypothyroid; hypoovarial; pituitary-hypothalamic disorders; adrenopathy.
   * iatrogenic (caused by drug administration, for example, insulin, glucocorticosteroids, neuroleptics etc.).
2. Compliance with a diet prescribed and monitored by the doctor to reduce body weight within 6 months before enrollment.
3. Participation in the lifestyle modification program within 6 months before enrollment.
4. Patients who quit smoking within 6 months before enrollment, or intending to quit smoking during the period of participation in the trial, as well as intending to begin smoking during the trial.
5. Uncontrolled arterial hypertension (patients with 1-3 degree AH, receiving no adequate antihypertensive therapy).
6. Type 1 and 2 diabetes mellitus.
7. Edema syndrome with various etiology (chronic cardiac failure, nephrotic syndrome, hepatic cirrhosis).
8. Circulatory failure, IIА degree and above.
9. Decompensated cardiovascular disease, liver, kidney or gastrointestinal tract disease, metabolic, respiratory, endocrine, hematologic disease, peripheral vessel disease or another medical state. Oncological disease.
10. Diseases and states, which, in the investigator's opinion, may prevent the patient from participating in the trial.
11. Past history of bulimia / non-drug anorexia.
12. Past history of any bariatric surgeries.
13. Lipoplasty underwent less then 1 year prior to screening visit, or cavitary surgery less then 6 months prior to screening visit.
14. Surgeries scheduled within 6 months.
15. Allergy to/intolerance of any of the drug components used during treatment.
16. Malabsorption syndrome, including congenial or acquired lactase or another disaccharidase insufficiency.
17. Administration of drugs specified as "Prohibited concomitant therapy", within 6 months before enrollment.
18. Pregnancy, breast-feeding, unwillingness to comply with contraception methods during the trial and within 30 days after completion of participation in the trial.
19. Drug and alcohol consumption (over 2 alc. units daily), mental diseases.
20. Legal incapacity or limited legal capacity.
21. Patients, who, in the investigator's opinion, will fail to observe the requirements during the trial or adhere to the studied drug administration procedure.
22. Participation in other clinical trials within 3 months before enrolment in this trial.
23. Presence of other factors, complicating the patient's participation in the trial (e.g., planned lengthy business and other trips).
24. A patient is a part of the center's research staff, taking a direct part in the trial, or an immediate family member of the investigator. Immediate family members are defined as spouses, parents, children or siblings, regardless of whether full blood or adopted.
25. The patient is employed with Scientific Production Firm Materia Medica Holding LLC, i.e. is the company's employee, part-time employee under contract, or appointed official in charge of the trial, or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - The State Educational institution of High Professional Training Kuban State Medical University of Ministry of Health Care and Social Development of the Russian Federation, Department of Clinical Pharmacology, Krasnodar
  - First Moscow State Medical University named after I.M. Sechenov/Endocrinology Faculty, Moscow
  - The State Budget Health Care institution of Moscow the City Clinical Hospital No. 11 of the Administration of Health Care of Moscow City, Moscow
  - Municipal Medical and Preventive institution "City Clinical Hospital No.10", Nizhny Novgorod
  - The State Budget Health Care institution of Nizhegorodskyi Region "Nizhegorodskaya Regional Clinical Hospital n.a. N.A.Semashko", Nizhny Novgorod
  - The State Educational institution of High Professional Training "Rostov State Medical University" of Ministry of Health Care and Social Development of the Russian Federation, Department of Endocrinology, Rostov-on-Don
  - St. Petersburg State Health Care institution "Municipal Hospital No.6", Saint Petersburg
  - St. Petersburg State Health Care institution "Municipal Hospital No.77 of Nevsky District", The City Diabetes Center, Saint Petersburg
  - The Federal State Health Care institution L.G. Sokolov Memorial Hospital No. 122 of the FMBA (Federal Medical and Biological Agency)., Saint Petersburg
  - The State Educational institution of High Professional Training "St. Petersburg State Medical University n.a. I.P. Pavlov of the Federal Agency for Health Care and Social Development", Faculty Surgery Board, Saint Petersburg
  - The State Educational institution of High Professional Training "St. Petersburg State Medical University n.a. I.P. Pavlov of the Federal Agency for Health Care and Social Development", Therapy Faculty Board, Saint Petersburg
  - St. Petersburg state Health Care institution "Saint Venerable Martyr Elizaveta Municipal Hospital", Saint Petersburg
  - St. Petersburg State Health Care institution "Consultative and Diagnostic Center No. 85", Diabetes Center, Saint Petersburg
  - The State Educational institution of High Professional Training "Bashkirsky State Medical University" of the Federal Agency for Health Care and Social Development, Department of Endocrinology, Ufa
  - The State Educational institution of High Professional Training "Volgograd State Medical University" of Ministry of Health Care and Social Development of the Russian Federation, Volgograd
  - The State Health Care institution "Voronezh Regional Clinical Consultative & Diagnostic Center", Voronezh
  - The State Health Care institution of Yaroslavl Region the Clinical Hospital, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dietressa | Placebo
Started | 164 | 167
Completed | 164 | 167
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietressa | Placebo | Total
Number analyzed (Participants) | 164 | 167 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.4) | 42.8 (11.6) | 43.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 139 | 277
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 164 | 167 | 331

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least 5% Weight Loss.
Description: Based on medical records.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
Participants | 80 | 62
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0352, Fisher Exact

2. Primary Outcome: Average Absolute Weight Change
Description: Based on medical records.
Time Frame: On baseline and after 24 weeks
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
kilogram
  Baseline | 104.7 (11.6) | 105.3 (11.4)
  After 24 weeks | 98.6 (12.7) | 101.3 (12.1)
  ∆ between baseline and after 24 weeks | 6.1 (5.3) | 4.0 (4.6)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Average Relative Weight Change
Description: Based on medical records.
Time Frame: On baseline and after 24 weeks
Population: ∆ between baseline and after 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of weight loss from baseline
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
percentage of weight loss from baseline | 5.9 (5.1) | 3.8 (4.4)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Patients With at Least 5% Weight Loss.
Description: Based on medical records.
Time Frame: On baseline and after 4, 8, 12, 16, 20, 24 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
Participants
  Baseline | 0 | 0
  After 4 weeks | 11 | 5
  After 8 weeks | 29 | 19
  After 12 weeks | 49 | 32
  After 16 weeks | 59 | 42
  After 20 weeks | 73 | 49
  After 24 weeks | 80 | 62
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Breslow-Day test p-value is 0.98

5. Secondary Outcome: Average Absolute Weight Change
Description: Based on medical records.
Time Frame: After 4, 8, 12, 16 and 20 weeks of treatment
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
kilogram
  Average absolute weight reduction after 4 weeks | 1.8 (2.2) | 1.3 (1.8)
  Average absolute weight reduction after 8 weeks | 2.9 (3.1) | 2.1 (2.6)
  Average absolute weight reduction after 12 weeks | 3.8 (3.9) | 2.8 (3.2)
  Average absolute weight reduction after 16 weeks | 4.7 (4.6) | 3.3 (3.7)
  Average absolute weight reduction after 20 weeks | 5.5 (4.9) | 3.7 (4.1)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0004, ANOVA — The p-value associated with "treatment*visit" interaction of changes from baseline to Week 4, 8, 12, 16 and 20 endpoint between Dietressa and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

6. Secondary Outcome: Average Relative Weight Change
Description: Based on medical records.
Time Frame: After 4, 8, 12, 16 and 20 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of weight loss from baseline
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
percentage of weight loss from baseline
  Average relative weight reduction after 4 weeks | 1.7 (2.1) | 1.3 (1.7)
  Average relative weight reduction after 8 weeks | 2.8 (2.9) | 2.0 (2.5)
  Average relative weight reduction after 12 weeks | 3.7 (3.7) | 2.7 (3.0)
  Average relative weight reduction after 16 weeks | 4.5 (4.4) | 3.2 (3.5)
  Average relative weight reduction after 20 weeks | 5.3 (4.8) | 3.5 (4.0)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; Test type: Superiority; p = 0.0004, ANOVA — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change in Waist Circumference, Waist Circumference/Hip Circumference.
Description: Based on medical records.
Time Frame: After 4, 12 and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
centimeter
  Change in waist circumference after 4 weeks | 2.2 (3.3) | 2.6 (3.5)
  Change in waist circumference after 12 weeks | 4.8 (5.2) | 4.7 (5.4)
  Change in waist circumference after 24 weeks | 6.9 (10.7) | 6.9 (6.1)
  Change in waist circumference/hip circumference after 4 weeks | 0.01 (0.03) | 0.01 (0.03)
  Change in waist circumference/hip circumference after 12 weeks | 0.01 (0.04) | 0.01 (0.05)
  Change in waist circumference/hip circumference after 24 weeks | 0.01 (0.04) | 0.01 (0.04)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; This analysis applies to rows with waist circumference data; Test type: Superiority; p = 0.67, ANOVA — The p-value associated with "treatment*visit" interaction of changes from baseline to Week 4, 12, and 24 endpoint between Dietressa and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction
Statistical Analysis 2: Comparison: Dietressa vs Placebo; This analysis applies to rows with hip circumference data; Test type: Superiority; p = 0.26, ANOVA — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Dynamics of the Quality of Life According to the SF-36 Questionnaire.
Description: Based on medical records. The short version of the SF-36 quality of life questionnaire is completed at visits 1, 2, 4, 7. The SF-36 questionnaire form consists of 11 sections, in each of which it is required to circle one number on each line. The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical activity score of the SF-36. Items 5-8 primarily contribute to the mental health score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement. The 'overall' estimate is the average change from baseline
Time Frame: On baseline and after 4, 12, 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dietressa | Placebo
Number analyzed (Participants) | 164 | 167
score on a scale
  Baseline Physical Health domain | 46.6 (8.1) | 47.3 (8.4)
  After 4 weeks Physical Health domain | 47.7 (7.8) | 49.0 (8.0)
  After 12 weeks Physical Health domain | 49.1 (7.6) | 49.7 (7.7)
  After 24 weeks Physical Health domain | 49.7 (6.8) | 50.9 (7.1)
  Baseline Mental Health domain | 44.7 (10.8) | 46.3 (9.7)
  After 4 weeks Mental Health domain | 48.2 (9.9) | 48.5 (9.3)
  After 12 weeks Mental Health domain | 48.3 (9.4) | 49.2 (8.9)
  After 24 weeks Mental Health domain | 49.2 (8.4) | 50.4 (8.3)
Statistical Analysis 1: Comparison: Dietressa vs Placebo; This analysis applies to rows with Physical Health domain data; Test type: Superiority; p = 0.40, ANOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Dietressa vs Placebo; This analysis applies to rows with Mental Health domain data; Test type: Superiority; p = 0.34, ANOVA — [p-value comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: During the study - 24 weeks.
Arm/Group | Dietressa | Placebo
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/167
Serious Adverse Events (participants affected / at risk) | 2/164 | 3/167
Other Adverse Events (participants affected / at risk) | 76/164 | 64/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietressa (N=164) | Placebo (N=167)
Membranous nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Gangrenous appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Closed fracture of the right leg and right foot as a result of a fall
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietressa (N=164) | Placebo (N=167)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) — Heartburn
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Viral respiratory tract infection (Infections and infestations) | 13 (13) | 8 (8)
Nail bed infection (Infections and infestations) | 1 (1) | 0 (0)
Candida Infection (Infections and infestations) | 1 (1) | 0 (0) — Thrush
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth pulpitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Abnormal glucose tolerance test results (Investigations) | 0 (0) | 2 (2)
Deviation from the ESR norm (Investigations) | 1 (1) | 0 (0)
Increased blood pressure (Investigations) | 1 (1) | 1 (1)
Increased ESR (Investigations) | 2 (2) | 1 (1)
Increased ALT (Investigations) | 2 (2) | 0 (0)
Increased AST (Investigations) | 1 (1) | 0 (0)
Increased blood glucose (Investigations) | 4 (4) | 2 (2)
Increased lymphocytes (Investigations) | 1 (1) | 0 (0)
Increase in LDL cholesterol (Investigations) | 1 (1) | 0 (0)
Increased monocytes (Investigations) | 1 (1) | 1 (1)
Increased platelets (Investigations) | 0 (0) | 2 (2)
Increased eosinophils (Investigations) | 0 (0) | 2 (2)
Increased red blood cells (Investigations) | 0 (0) | 2 (2)
Elevated LDL (Investigations) | 1 (1) | 0 (0)
Elevated triglycerides (Investigations) | 0 (0) | 2 (2)
Decreased serum creatinine levels (Investigations) | 0 (0) | 1 (1)
Decreased platelets (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 1 (1)
Increased LDL to HDL ratio (Investigations) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyslipidemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Impaired fasting glycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type II diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia, unspecified (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Degenerative changes in the thoracic spine
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Lumbago
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Deforming osteoarthritis
Subchondral bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Increased activity (Nervous system disorders) | 0 (0) | 1 (1) — Psychomotor hyperactivity
Retinal dystrophy (Eye disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bartholin's gland cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstrual disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Tibial vein thrombosis
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Increased body temperature (General disorders) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 18 (18) | 10 (10)
Depression, worsening (Psychiatric disorders) | 12 (12) | 13 (13)
Feeling of elation (Psychiatric disorders) | 1 (1) | 1 (1) — Euphoric mood
Increased anxiety (Psychiatric disorders) | 32 (32) | 36 (36)
Bruised toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes